CLINICAL TRIAL: NCT00224588
Title: Effects of Peri Operative Administration of Ketamine on Long Term Post Thoracotomy Pain
Brief Title: KETOR: Effects of Peri Operative Administration of Ketamine on Long Term Post Thoracotomy Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Direction Régionale de la Recherche Clinique D'ILE DE FRANCE (Unknown); Clinical Research Unit (Ambiguous); European Georges Pompidou Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P990911; CRC99029
Record Dates: First submitted 2005-09-16; First posted 2005-09-23 (Estimated); Last update posted 2006-04-13 (Estimated); Status verified 2005-09

CONDITIONS: Ketamine; Chronic Post Thoracotomy Pain; Thoracotomy; Pain; Neuralgia
Keywords: Ketamine; Chronic post thoracotomy pain; NMDA; Post operative
MeSH Terms: conditions — Pain; Neuralgia | interventions — Ketamine

INTERVENTIONS:
Drug: Ketamine (or placebo : isotonic saline solution)

SUMMARY:
We assessed the effects of the N Methyl aspartate receptor antagonist Ketamine on long-term post thoracotomy pain. We hypothesized that ketamine could prevent supersensitization of the central nervous system involved in this chronic neuropathic pain.

DETAILED DESCRIPTION:
In this clinical, randomized prospective study, peri operative administration of ketamine was compared to placebo on long term post thoracotomy pain after a 2 months follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for thoracotomy or pneumectomy

Exclusion Criteria:

-

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80
Dates: Start 2003-01; Study Completion 2005-05

PRIMARY OUTCOMES:
Long term (2 months) post thoracotomy pain was assessed using a french equivalent of the Mc Gill Pain score and pain area measurements in both groups

SECONDARY OUTCOMES:
Analogic pain scores at rest and after coughing

CONTACTS AND LOCATIONS:
Overall Officials: Thierry GUENOUN, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Georges Pompidou European Hospital, Paris, Île-de-France Region, France

REFERENCES:
- [Background] Frappier J, Guenoun T, Journois D, Philippe H, Aka E, Cadi P, Silleran-Chassany J, Safran D. Airway management using the intubating laryngeal mask airway for the morbidly obese patient. Anesth Analg. 2003 May;96(5):1510-1515. doi: 10.1213/01.ANE.0000057003.91393.3C. PMID 12707159